CLINICAL TRIAL: NCT05469659
Title: Effect of Tofogliflozin on Urine Albumin-to-Creatinine Ratio Compared to Metformin Hydrochloride in Diabetic Kidney Disease
Brief Title: Effect of Tofogliflozin on UACR Compared to Metformin Hydrochloride in Diabetic Kidney Disease (TRUTH-DKD)
Acronym: TRUTH-DKD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shinshu University (Other)
Collaborators: Kowa Company, Ltd. (Industry)
Responsible Party: Principal Investigator, Koichiro Kuwahara, MD, PhD, Professor, Shinshu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-02; jRCTs031210339 (Registry Identifier: jRCT)
Record Dates: First submitted 2022-07-15; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: T2DM (Type 2 Diabetes Mellitus); Metformin; SGLT2-Inhibitors
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 6-((4-ethylphenyl)methyl)-3',4',5',6'-tetrahydro-6'-(hydroxymethyl)spiro(isobenzofuran-1(3H),2'-(2H)pyran)-3',4',5'-triol; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tofogliflozin (Experimental)
  Interventions: Drug: Tofogliflozin
- Metformin (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Tofogliflozin — Tofogliflozin 20 mg is orally administered once daily for 104 weeks before or after breakfast.
  Arms: Tofogliflozin
Drug: Metformin — Metformin is started at 500 mg daily and orally administered in 2 to 3 divided doses immediately before or after meals. The dose during the maintenance period is determined by observing the effect, but is usually 750 to 1,500 mg daily. Metformin is orally administered for 104 weeks throughout post-start period. The dose may be adjusted according to the patient's condition, but the maximum daily dose should be 2,250 mg.
  Arms: Metformin

SUMMARY:
This multicenter, randomized, open-label, controlled study will assess the efficacy of the SGLT2 inhibitor tofogliflozin on Urine Albumin-to-Creatinine Ratio (UACR) compared to metformin in patients with type 2 diabetes with chronic kidney disease (CKD).

DETAILED DESCRIPTION:
Eligible participants will be randomly assigned (1:1) to tofogliflozin or metformin with stratification based on UACR (<300 mg/gCr，≧300mg/gCr), an estimated glomerular filtration rate (eGFR) (<60mL/min/1.73m2, ≧60 mL/min/1.73m2), and age (<65 years old, ≧65 years old). The primary end point is change in urine albumin-to-creatinine ratio (UACR) from baseline after 52 weeks treatment. Changes in eGFR, HbA1c, body weight, systolic blood pressure, diastolic blood pressure, total serum proteins, serum albumin, uric acid, hematocrit, hemoglobin, red blood cell count, pulse rate, triglyceride, low-density lipoprotein, high-density lipoprotein and albuminuria class transition rate will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients
* Patients aged 20 years or older at the time of obtaining consent
* Patients with HbA1c 6.5 or more and 9.0% or less within 13 weeks before obtaining consent (evaluated by test values after 4 weeks or more without taking SGLT2 inhibitor / metformin)
* Patients who have been judged by their doctor to need a diabetic drug when they are first seen, or who have already taken a diabetic drug and have decided that it is necessary to add one diabetic drug.
* Patients who have been receiving RAS inhibitors (ARB, ARNI, ACE inhibitors, direct renin inhibitors) for 4 weeks or longer
* Patients with eGFR of 30 or more (mL / min / 1.73m2) within 13 weeks before obtaining consent (evaluated by test values after 4 weeks or more without taking SGLT2 inhibitor / metformin)
* Patients with urinary albumin / creatinine ratio (UACR) of 30 or more and less than 2000 (mg / gCr) (4 weeks or more without taking SGLT2 inhibitor / metformin) within 13 weeks before obtaining consent Evaluate by inspection value)
* Patients for whom written consent was obtained based on the patient's free will after receiving sufficient explanation for participation in this study

Exclusion Criteria:

* Patients receiving treatment with SGLT2 inhibitor or metformin within 13 weeks before obtaining consent
* Dialysis patient
* Patients with a history of severe hypoglycemia
* Patients with hypersensitivity to SGLT2 inhibitor or metformin
* Pregnant women, lactating patients, and patients who wish to raise children
* Patients with BMI of 35 kg / m2 or more based on the latest measured values within 13 weeks before obtaining consent
* Patients who are contraindicated for the study drug
* Other patients who the attending physician deems inappropriate as a subject

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Urine albumin-to-creatinine ratio (UACR) | Up to 52 weeks
  Change from baseline in urine albumin-to-creatinine ratio (UACR) after 52 weeks treatment.

SECONDARY OUTCOMES:
Urine albumin-to-creatinine ratio (UACR) | Up to 26 and 104 weeks
  Change from baseline in urine albumin-to-creatinine ratio (UACR) after 26 and 104 weeks treatment.
Urine albumin-to-creatinine ratio (UACR) | Up to 26, 52 and 104 weeks
  Change rates from baseline in urine albumin-to-creatinine ratio (UACR) after 26, 52 and 104weeks treatment.
Change slope in eGFR | Up to 52 and 104 weeks
  Change slope in eGFR
HbA1c | Up to 52 and 104 weeks
  Change in HbA1c
Body weight | Up to 52 and 104 weeks
  Changes in body weight
Systolic / diastolic blood pressure | Up to 52 and 104 weeks
  Changes in systolic / diastolic blood pressure
Total serum proteins | Up to 52 and 104 weeks
  Changes in total serum proteins
Serum albumin | Up to 52 and 104 weeks
  Changes in serum albumin
Uric acid | Up to 52 and 104 weeks
  Changes in uric acid
Hematocrit | Up to 52 and 104 weeks
  Changes in hematocrit
Hemoglobin | Up to 52 and 104 weeks
  Changes in hemoglobin
Red blood cell count | Up to 52 and 104 weeks
  Changes in red blood cell count
Pulse rate | Up to 52 and 104 weeks
  Changes in pulse rate
Triglyceride | Up to 52 and 104 weeks
  Changes in triglyceride
Low-density lipoprotein | Up to 52 and 104 weeks
  Changes in low-density lipoprotein
High-density lipoprotein | Up to 52 and 104 weeks
  Changes in high-density lipoprotein
Albuminuria class | Up to 104 weeks
  Transition of albuminuria class

CONTACTS AND LOCATIONS:
Overall Officials: Koichiro Kuwahara, MD, PhD, Study Chair — Shinshu University School of Medicine
Locations (1):
- Shinshu University, Matsumoto, Nagano, Japan

REFERENCES:
- [Derived] Kimura K, Takagi Y, Harada M, Ueda S, Minamisawa M, Sonoda K, Oiwa A, Yazaki Y, Sakurai S, Tomita T, Kaneko K, Yamamoto K, Takama N, Momose S, Inobe Y, Nogi K, Koshikawa M, Misawa T, Kasai T, Tsutsui H, Watanabe N, Yamazaki K, Miyamoto T, Midorikawa T, Usui T, Saigusa T, Motoki H, Saito Y, Kamijo Y, Komatsu M, Kuwahara K. Effect of Tofogliflozin on Urinary Albumin-to-Creatinine Ratio vs. Metformin in Diabetic Kidney Disease: Rationale and Study Protocol of the TRUTH-DKD Trial. Diabetes Ther. 2025 Nov 18. doi: 10.1007/s13300-025-01822-8. Online ahead of print. PMID 41252113
- [Derived] El-Damanawi R, Stanley IK, Staatz C, Pascoe EM, Craig JC, Johnson DW, Mallett AJ, Hawley CM, Milanzi E, Hiemstra TF, Viecelli AK. Metformin for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2024 Jun 4;6(6):CD013414. doi: 10.1002/14651858.CD013414.pub2. PMID 38837240